CLINICAL TRIAL: NCT06505707
Title: The Effect of Health Seeking Behavior Training Based on Motivational Interviewing Techniques on Health Seeking Behavior, Illness Self-Management and Anxiety in Immigrant Elderly Women With Chronic Disease: A Randomized Controlled Trial
Brief Title: The Effect of Motivational Interviewing-Based Health Behavior Training in Chronically Ill Migrant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Pinar Harmanci, Assistant Professor, Kahramanmaraş İstiklal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstiklalU-Harmanci-001
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Motivational Interviewing; Health Care Seeking Behavior; Migrants; Women
Keywords: Elderly; Self Efficacy; Anxiety
MeSH Terms: conditions — Patient Acceptance of Health Care; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Seeking Behavior Training Based on Motivational Interviewing Techniques (Experimental): The "Migrant Elderly Women with Chronic Diseases" in the intervention group, who will receive Health Seeking Behavior Training based on Motivational Interviewing Techniques, will be divided into four groups (the researcher conducting the intervention will interview the individuals in the 4 groups individually for 4 days). The interviews will be conducted 4 days a week (Monday, Tuesday, Thursday and Friday) and the Health Seeking Behavior Training based on Motivational Interviewing Techniques, which lasts 4 weeks and each session is approximately 30-35 minutes, will be applied face-to-face.
  Interventions: Behavioral: Health Seeking Behavior Training Based on Motivational Interviewing Techniques
- Control group (No Intervention): There will be no intervention for individuals in this group.

INTERVENTIONS:
Behavioral: Health Seeking Behavior Training Based on Motivational Interviewing Techniques — The Effect of Health Seeking Behavior Training Based on Motivational Interviewing Techniques on Health Seeking Behavior, Illness Self-Management and Anxiety in Migrant Elderly Women with Chronic Diseases.
  Arms: Health Seeking Behavior Training Based on Motivational Interviewing Techniques

SUMMARY:
This randomized controlled experimental study will be conducted to investigate the effect of health seeking behavior training based on motivational interviewing techniques on health seeking behaviors, illness self-management and anxiety in migrant elderly women with chronic illness.

Hypotheses of the Study H11: Health-seeking behaviors training based on motivational interviewing techniques with migrant elderly women with chronic diseases will improve individuals' correct health-seeking behaviors.

H12: Health seeking behaviors training based on motivational interviewing techniques with migrant elderly women with chronic diseases will increase individuals' disease self-management.

H13: Health-seeking behaviors training based on motivational interviewing techniques with migrant elderly women with chronic diseases will reduce the anxiety level of individuals.

In the study, there will be an intervention group in which health-seeking behavior training based on motivational interviewing techniques will be applied and a control group in which no intervention will be applied.

The "Migrant Elderly Women with Chronic Diseases" in the intervention group, who will receive Health Seeking Behavior Training based on Motivational Interviewing Techniques, will be divided into four groups (the researcher conducting the intervention will interview the individuals in the 4 groups individually for 4 days). The interviews will be conducted 4 days a week (Monday, Tuesday, Thursday and Friday) and the Health Seeking Behavior Training Based on Motivational Interviewing Techniques, which lasts 4 weeks and each session is approximately 30-35 minutes, will be applied face-to-face.

DETAILED DESCRIPTION:
''Migrant Elderly Women with Chronic Diseases'' who constitute the sample of the study will be informed about the Health Seeking Behavior Training based on Motivational Interviewing Techniques by obtaining the necessary permissions. After the intervention group and control group are determined by simple randomization method, pre-tests will be applied to both groups through face-to-face interviews. For the individuals in the intervention group, the days on which the Health Seeking Behavior Training Based on Motivational Interviewing Techniques will be implemented will be determined. The "Migrant Elderly Women with Chronic Diseases" in the intervention group who will receive Health Seeking Behavior Training based on Motivational Interviewing Techniques will be divided into four groups (the researcher who will conduct the application will interview the individuals in the 4 groups individually for 4 days). The interviews will be conducted 4 days a week (Monday, Tuesday, Thursday and Friday), lasting 4 weeks and each session will last approximately 30-35 minutes. Individuals who will come to the face-to-face training and belong to the intervention group divided into four will be called by the researcher for the training and called to a room with a therapeutic environment at the university. In addition, interviews will be continued by providing a therapeutic environment. The researcher will conduct interviews with each group on the days and times they have jointly planned. Thus, face-to-face practice will be carried out with a group every day. After the completion of the Health Seeking Behavior Training based on Motivational Interviewing Techniques, post-tests will be applied to the intervention and control groups through face-to-face interviews.

In the control group, pre-tests will be collected and no intervention will be made. For the post-test, the patients will be interviewed face-to-face on the agreed appointment date and post-test data will be collected in line with the data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* Migrant older women aged 65 years and older with chronic diseases,
* Immigrant women who have been living in Turkey for at least six months and who may or may not have acquired citizenship,
* Women who have no communication problems and who volunteered to be included in the study

Exclusion Criteria:

* Women with dementia, Alzheimer's disease and diagnosed mental illness with a mini-mental test score below 24

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Health Seeking Behavior Scale | 0 weeks
  It was developed by Kıraç and Öztürk in 2019 to assess individuals' health seeking behavior. The scale consists of 12 questions and three sub-dimensions: online health seeking behavior, professional health seeking behavior and traditional health seeking behavior. The score to be obtained from the scale varies between 12-60 and the scores obtained are divided by the number of scale items and an average between 1-5 points is obtained. The increase in the scores obtained from the total scale and its sub-dimensions indicates that the health seeking behavior of the individual increases.
Health Seeking Behavior Scale | 4 weeks
  It was developed by Kıraç and Öztürk in 2019 to assess individuals' health seeking behavior. The scale consists of 12 questions and three sub-dimensions: online health seeking behavior, professional health seeking behavior and traditional health seeking behavior. The score to be obtained from the scale varies between 12-60 and the scores obtained are divided by the number of scale items and an average between 1-5 points is obtained. The increase in the scores obtained from the total scale and its sub-dimensions indicates that the health seeking behavior of the individual increases.
Health Anxiety Scale | 0 weeks
  The scale developed by Salkovskis et al. in 2002 is a self-report scale consisting of 18 items. The Turkish validity and reliability of the scale was conducted by Aydemir et al. in 2013. The scale consists of 18 items. Fourteen items of the scale consist of statements containing quadruple responses questioning the mental status of the patients. The total score that can be obtained from the scale varies between 0 and 54 points. A high score on the scale indicates a high level of health anxiety.
Health Anxiety Scale | 4 weeks
  The scale developed by Salkovskis et al. in 2002 is a self-report scale consisting of 18 items. The Turkish validity and reliability of the scale was conducted by Aydemir et al. in 2013. The scale consists of 18 items. Fourteen items of the scale consist of statements containing quadruple responses questioning the mental status of the patients. The total score that can be obtained from the scale varies between 0 and 54 points. A high score on the scale indicates a high level of health anxiety.
Chronic Disease Self-Management Scale | 0 weeks
  The Turkish validity and reliability of the scale developed by Ngai et al. in 2020 was conducted by Öztürk et al. in 2021. The Turkish version of the scale consists of 23 items and 4 sub-dimensions. The sub-dimensions of the scale are self-stigmatization, coping with stigmatization, health care effectiveness and treatment compliance. The scale items are in a 5-point Likert scale and are scored between 5 and 5.
Chronic Disease Self-Management Scale | 4 weeks
  The Turkish validity and reliability of the scale developed by Ngai et al. in 2020 was conducted by Öztürk et al. in 2021. The Turkish version of the scale consists of 23 items and 4 sub-dimensions. The sub-dimensions of the scale are self-stigmatization, coping with stigmatization, health care effectiveness and treatment compliance. The scale items are in a 5-point Likert scale and are scored between 5 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin SAZAK, Principal Investigator — Kahramanmaraş İstiklal University